CLINICAL TRIAL: NCT07152119
Title: Korean Post Marketing Surveillance for Litfulo Capsule
Brief Title: A Study to Learn About Litfulo Capsule in People With Severe Alopecia Areata in Routine Clinical Practice.
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7981084
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Severe Alopecia Areata
Keywords: Litfulo; Litfulo capsule; Ritlecitinib tosylate
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe alopecia areata.: Determined to start treatment with Litfulo Capsule according to the approved indications of the medicinal product.
  Interventions: Drug: Litfulo

INTERVENTIONS:
Drug: Litfulo — as provided in real world practice.
  Other Names: Ritlecitinib tosylate (ATC code: L04AF08)

SUMMARY:
The purpose of this observation study is to learn about the safety and effects of the study medicine (called Litfulo) for the potential treatment of Severe Alopecia Areata.

DETAILED DESCRIPTION:
To evaluate the safety of Litfulo Capsule after marketing, with regard to the following clauses in routine clinical practice.

* Adverse Events (AEs)/ Adverse Drug Reactions (ADRs)
* Unexpected Adverse Events (AEs)/ADRs that have not been reflected in the approved drug label
* Serious Adverse Events (SAEs)/Serious Adverse Drug Reaction (SADRs)
* Adverse Event of Special Interest(AESI)

  * Serious Infections, defined as any infection (viral, bacterial, and fungal) requiring parenteral antimicrobial therapy or hospitalization for treatment or meeting other criteria that require the infection to be classified as serious adverse event
  * Opportunistic infections and Herpes Zoster
  * Malignancy

ELIGIBILITY:
Inclusion Criteria:

Patients with severe alopecia areata who have been determined to start treatment with Litfulo Capsule according to the approved indications of the medicinal product Treatment of severe alopecia areata in adults and adolescents 12 years or older Evidence of a personally signed and dated informed consent document indicating that the patient or their parent(s)/legal guardian, if applicable, have been informed of all pertinent aspects of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe alopecia areata
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2030-03-23 (Estimated); Study Completion 2030-03-23 (Estimated)

PRIMARY OUTCOMES:
Frequency and proportion of AEs/ADRs | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Frequency and proportion of unexpected AEs/ADRs | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Frequency and proportion of SAEs/SADRs | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Frequency and proportion of AESI | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)

SECONDARY OUTCOMES:
Proportion of patients achieving Severity of Alopecia Tool (SALT) ≤20 score at Weeks 24 and 48 | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Proportion of patients achieving SALT ≤10 score at Weeks 24 and 48 | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Proportion of patients achieving 50% or above improvement in SALT score from baseline (SALT 50) at Weeks 24 and 48 | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)
Proportion of patients achieving 75% or above improvement in SALT score from baseline (SALT 75) at Weeks 24 and 48 | 24 weeks (Regular surveillance), 48 weeks (Long-term surveillance)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981084